CLINICAL TRIAL: NCT00504101
Title: Phase I Clinical Trial of Dose Escalated Bortezomib + ATO (Arsenic Trioxide) + Melphalan as a Conditioning Regimen for Multiple Myeloma
Brief Title: Bortezomib, Arsenic Trioxide, and Melphalan in Treating Patients Undergoing an Autologous Stem Cell Transplant For Multiple Myeloma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Temporarily closed to accrual pending availablity of drug.
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20070104; SCCC-2006071 (Other: University of Miami Sylvester Comprehensive Cancer Center)
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Arsenic Trioxide; Bortezomib; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Arsenic trioxide — Arsenic Trioxide will be given on day -6, -5, -4,-3,-2 (total of 5 doses). The dose of Arsenic trioxide (ATO) is 0.25 mg/m2.
  Other Names: ATO (As2O3)
Drug: Bortezomib — Bortezomib will be given on day -6, -4, -2 (total 3 doses) beginning at a dose of 0.8 mg/m2 each day of therapy.
  Other Names: Velcade; PS-341
Drug: Melphalan — Melphalan will be given at 200 mg/m2 on day -2 (1 dose only)
  Other Names: L-PAM; L-phenylalanine mustard; L-sarcolysin; Alkeran
Biological: Autologous hematopoietic stem cell transplantation — On day 0 a minimal of 2 x 106 CD 34 cells/kg will be infused by central catheter according to institutional standards.

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as arsenic trioxide and melphalan, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving high-dose combination chemotherapy together with bortezomib may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of bortezomib when given together with arsenic trioxide and melphalan in treating patients undergoing an autologous stem cell transplant for multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate toxicity of a conditioning treatment regimen comprising bortezomib, arsenic trioxide, and melphalan.

Secondary

* Evaluate response and overall survival.
* Determine what correlative laboratory and clinical parameters, if any, are associated with efficacy (e.g., serum arsenic trioxide intracellular glutathione depletion, gene profiling of myeloma cells).

OUTLINE: This is a dose-escalation study of bortezomib.

* Conditioning regimen: Bortezomib will be given on days -6, -4, and -2, arsenic trioxide will be given on days -6, -5, -4, -3, and -2 (total of 5 doses), and melphalan will be given on day -2.
* Stem cell infusion: On day 0 a minimum of autologous 2 x 10^6 CD34 cells/kg will be infused by central catheter.

After completion of study therapy, patients are followed periodically for at least 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Confirmed diagnosis of multiple myeloma (M-protein by serum protein electrophoresis or urine protein electrophoresis) and either bone marrow biopsy and aspirate demonstrating a plasma cell count > 10% or biopsy of a bone or soft tissue mass demonstrating a plasmacytoma

  * Demonstration of an indication for therapy based on symptoms (e.g., boney pain), hypercalcemia, anemia, renal insufficiency, symptomatic plasmacytomas, multiple boney lytic lesions, etc
  * Stable disease or has achieved a partial remission or complete remission to pre-transplant cyto-reductive therapy
  * Primary refractory disease (no response to therapy but stable) is permitted
* Candidate for high-dose chemotherapy with autologous stem cell transplantation based on stabilization of disease with preparative chemotherapy (regardless of the specific agents)
* A minimum of 2 x 10^6 CD34+ cells/kg must be collected prior to proceeding to transplant

Exclusion criteria:

* Evidence of active plasma cell leukemia
* Relapsed refractory disease (patients who have achieved at least a partial response [PR] to previous therapy and are now refractory [have not achieved a PR to subsequent therapy])
* Progressive disease on their last therapy

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Karnofsky performance status 60-100%
* Creatinine < 3.0 mg/dL
* AST and ALT <2.5 times upper limit of normal
* Total bilirubin < 3 mg/dL
* WBC ≥ 2,000/mm³
* Platelet count ≥ 50,000/mm³
* If abnormal hematologic function is attributable to bone marrow infiltration by multiple myeloma, the principal investigator will decide on a case-by-case basis if the patient's bone marrow reserve is appropriate for this study
* Females of childbearing potential must have a negative serum pregnancy test prior to enrollment on the study and must use an effective barrier method while on the study
* Ejection fraction > 40% and no history of uncontrolled ischemic heart disease or congestive heart failure
* No evidence of cardiac amyloidosis by echocardiogram
* DLCO and FEV_1 ≥ 50%

Exclusion criteria:

* Active peripheral neuropathy ≥ grade 2
* Recurrent supraventricular arrhythmia or any type of sustained ventricular arrhythmia or conduction block (e.g., A-V block grade II or III, left bundle branch block)
* Known HIV infection
* Pregnant or lactating women
* Underlying medical condition that could be aggravated by the treatment or life-threatening disease unrelated to myeloma as evaluated by the enrolling physician
* History of second malignancy within the past 3 years and not in complete remission from that malignancy, excluding adequately treated basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or local prostate cancer
* History of preexisting neurological disorders (grade 2 or higher by the NCI Common Toxicity Criteria, in particular seizure disorders)

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* Previous radiation therapy for palliation of cord compression or pathologic fractures is permitted provided last dose is given 14 days prior to initiation of chemotherapy
* Subjects with radiographic evidence of lytic bone disease receiving concomitant bisphosphonate therapy may be enrolled

  * Bisphosphonates should be held at least 1 week prior to the transplant but continuing bisphosphonates after day +60 is at the discretion of the treating physician

Exclusion criteria:

* Previous autologous or allogeneic transplantation
* Other investigational or experimental drug or therapy while on the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Evaluate toxicity of the conditioning treatment regimen. | 3 ¼ years

SECONDARY OUTCOMES:
Evaluate response and overall survival (OS). | 3 ¼ years
Determine what correlative laboratory and clinical parameters, if any, are associated with efficacy | 3 ¼ years

CONTACTS AND LOCATIONS:
Overall Officials: Mark S. Goodman, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida, United States